CLINICAL TRIAL: NCT01217710
Title: Next Generation Technology for Chronic Care Self Management
Brief Title: Promoting Physical Activity in Chronic Obstructive Pulmonary Disease (COPD) Through New Technology and Health Coaching
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Roberto P. Benzo, Consultant Pulmonary and Critical Care Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-001171; 2R44AG029087-02A1 (NIH)
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Physical Activity
Keywords: Chronic Obstructive Pulmonary Disease; Physical Activity; Self Management; Exercise; Technology; Motivational Interviewing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Activity monitor/smartphone health coaching — Initial health coaching at enrollment will involve the collaborative creation of an action plan with personally relevant, specific actions for increasing physical activity. The short term goals will be rated for self-efficacy and modified to maximize likelihood of success. Health coaches will discuss important mediators of physical activity (e.g., self-efficacy, enjoyment, social support, problem-solving). Weekly coaching calls will involve discussion of progress toward goals and problem-solving of barriers utilizing a motivational interviewing approach. Motivational messages will also be developed and sent daily to participants via the smartphone. These messages will indicate the percentage of steps related to their daily goal.

SUMMARY:
The objective of this project is to validate the proposed smartphone-based activity monitor and to test its use for Motivational Interviewing based counseling for physical activity in Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 40 years and older
* Current or former smoker of at least 10 pack-years
* Diagnosis of GOLD stage II to IV COPD as documented by pulmonary function testing (FEV1 (Forced expiratory volume in 1 second) <80 percent predicted, FEV1/FVC(Forced vital capacity)<0.71)
* Able to walk independently or with a walking aid (e.g. wheeled walker, cane, standard walker)

Exclusion Criteria:

* Unable to walk without assistance of another person
* Patients with a high likelihood of being lost to follow-up or contact (patients with active chemical dependency), are planning to move out of the state, are not living in the healthcare area.
* Patients with an inability to provide good data or follow commands (patients who are disoriented, have a severe neurologic or psychiatric condition).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Validity of activity monitor/smartphone to accurately measure and record physical activity of COPD patients | 3 months
  Conduct tests to evaluate the activity monitor/smartphone system's ability to capture physical activity for COPD patients in comparison with the gold standard device in the field. The average number of steps and minutes per day spent in physical activities recorded by the experimental device will be compared to the gold standard device.

SECONDARY OUTCOMES:
Determine the feasibility of using the smartphone/activity monitoring technology for motivational interviewing based counseling . | 3 months
  Investigators will test the usability of the smartphone diary for chronic disease self-management health coaching. Several measures of the usability of the diary will be collected.
Determine the effectiveness of smartphone/activity monitor plus the motivational interviewing based coaching to increase physical activity, improve quality of life or palliate symptoms . | 3 months
  Several measures will be collected,Physical Activity Level (total energy expenditure/resting metabolic rate), steps, quality of life, self efficacy and also a qualitative feedback .

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, M.D., MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States